CLINICAL TRIAL: NCT00320489
Title: A Randomized, Open-label Study Comparing the Effects of Olanzapine Pamoate Depot With Oral Olanzapine on Treatment Outcomes in Outpatients With Schizophrenia
Brief Title: Olanzapine Pamoate Depot Versus Oral Olanzapine on Treatment Outcomes in Outpatients With Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6390; F1D-MC-HGLQ (Other: Eli Lilly and Company)
Record Dates: First submitted 2006-04-28; First posted 2006-05-03 (Estimated); Results first posted 2010-10-22 (Estimated); Last update posted 2012-01-23 (Estimated); Status verified 2012-01

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Olanzapine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Olanzapine Pamoate Depot (Experimental): Olanzapine pamoate depot
  Interventions: Drug: olanzapine pamoate depot
- Olanzapine (Active Comparator): Oral olanzapine
  Interventions: Drug: olanzapine

INTERVENTIONS:
Drug: olanzapine — 10 milligrams (mg), oral tablets, once daily for 4 weeks followed by 5-20 mg flexible dosing, oral tablets, once daily, for 100 weeks, for a total treatment duration of 104 weeks.
  Other Names: LY170053; Zyprexa
  Arms: Olanzapine
Drug: olanzapine pamoate depot — 405 milligrams (mg), intramuscular injection, followed 4 weeks later by 150-405 mg flexible dosing, intramuscular injection, every 4 weeks thereafter for 96 weeks, for a total treatment duration of 104 weeks.
  Arms: Olanzapine Pamoate Depot

SUMMARY:
To compare the health outcome of patients with schizophrenia, who are at risk for relapse, when treated with a long acting injection form of olanzapine versus treatment with oral olanzapine.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of schizophrenia
* Must be an outpatient (not requiring hospitalization) now and for at least the past 8 weeks.
* Disease symptoms must meet a certain range as assessed by the clinician.
* Patient has experienced at least two episodes of clinical worsening of their condition. This could mean admission to a hospital or an emergency room visit. This could mean that a new medication was added, medication dose was increased, or medication was switched in order to better control symptoms of the condition.
* The patient must have an unsatisfactory response to their current medication or be experiencing negative effects of their current medication or not always take their current medication so that a change in current medication is desired.

Exclusion Criteria:

* Patients who are actively suicidal.
* Patients who are pregnant or nursing.
* Patients who have stopped past treatment with olanzapine because of adverse events, are treatment resistant or allergic to olanzapine, or have a condition which would prevent use of a long acting form of olanzapine.
* Patients with uncorrected narrow-angle glaucoma, seizures, uncontrolled diabetes, certain diseases of the liver, uncontrolled thyroid condition or other serious or unstable illness.
* Patients with Parkinson's disease, psychosis related to dementia or other related disorders.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 524 (Actual)
Dates: Start 2006-04; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT- 5 hours, EST), Study Director — Eli Lilly and Company
Locations (49):
- United States (13):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Escondido, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., National City, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Orange, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Diego, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Washington D.C., District of Columbia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Honolulu, Hawaii
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chicago, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cedarhurst, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Staten Island, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Canton, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Allentown, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Philadelphia, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., West Chester, Pennsylvania
- Argentina (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Banfield
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Buenos Aires
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mendoza
- Brazil (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pelotas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rio de Janeiro
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., São Paulo
- Canada (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Calgary, Alberta
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Winnipeg, Manitoba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Burlington, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chatham, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Greater Sudbury, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Montreal, Quebec
- France (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dijon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dole
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., La Seyne-sur-Mer
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Limoges
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Strasbourg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toulon
- Greece (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chaïdári
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Haidari, Athens
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Thessaloniki
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tripoli
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lisbon, Portugal
- Puerto Rico (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cabo Rojo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Caguas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mayagüez
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rio Piedras
- Romania (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bucharest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Iași
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Târgu Mureş
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bratislava, Slovakia
- Spain (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Alzira
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barcelona
- Taiwan (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hua-Lian County
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taipei
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taoyuan

REFERENCES:
- [Derived] Atkins S, Detke HC, McDonnell DP, Case MG, Wang S. A pooled analysis of injection site-related adverse events in patients with schizophrenia treated with olanzapine long-acting injection. BMC Psychiatry. 2014 Jan 14;14:7. doi: 10.1186/1471-244X-14-7. PMID 24423017
- [Derived] Peuskens J, Porsdal V, Pecenak J, Handest P, D'yachkova Y, Brousil R, Deberdt W. Schizophrenia symptoms and functioning in patients receiving long-term treatment with olanzapine long-acting injection formulation: a pooled analysis. BMC Psychiatry. 2012 Aug 31;12:130. doi: 10.1186/1471-244X-12-130. PMID 22935168
- [Derived] McDonnell DP, Detke HC, Bergstrom RF, Kothare P, Johnson J, Stickelmeyer M, Sanchez-Felix MV, Sorsaburu S, Mitchell MI. Post-injection delirium/sedation syndrome in patients with schizophrenia treated with olanzapine long-acting injection, II: investigations of mechanism. BMC Psychiatry. 2010 Jun 10;10:45. doi: 10.1186/1471-244X-10-45. PMID 20537130
- [Derived] Detke HC, McDonnell DP, Brunner E, Zhao F, Sorsaburu S, Stefaniak VJ, Corya SA. Post-injection delirium/sedation syndrome in patients with schizophrenia treated with olanzapine long-acting injection, I: analysis of cases. BMC Psychiatry. 2010 Jun 10;10:43. doi: 10.1186/1471-244X-10-43. PMID 20537128
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Olanzapine Pamoate Depot: 405 mg, intramuscular injection, followed 4 weeks later by 150-405 mg flexible dosing, intramuscular injection, every 4 weeks thereafter for 96 weeks, for a total treatment duration of 104 weeks.
- Oral Olanzapine: 10 mg, oral tablets, once daily for 4 weeks followed by 5-20 mg flexible dosing, oral tablets, once daily, for 100 weeks, for a total treatment duration of 104 weeks.
Period: Overall Study
Arm/Group | Olanzapine Pamoate Depot | Oral Olanzapine
Started | 264 | 260
Completed | 119 | 124
Not Completed | 145 | 136
Not completed — Adverse Event | 26 | 25
Not completed — Clinical Relapse | 26 | 20
Not completed — Death | 0 | 2
Not completed — Entry Criteria Exclusion | 2 | 4
Not completed — Lack of Efficacy | 16 | 7
Not completed — Lost to Follow-up | 21 | 22
Not completed — Physician Decision | 8 | 8
Not completed — Protocol Violation | 4 | 4
Not completed — Sponsor Decision | 3 | 3
Not completed — Withdrawal by Subject | 39 | 41

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Olanzapine Pamoate Depot | Oral Olanzapine | Total
Number analyzed (Participants) | 264 | 260 | 524
Age Continuous [Mean (Standard Deviation); unit: years] | 41.70 (10.92) | 40.12 (10.84) | 40.92 (10.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 89 | 83 | 172
  Male | 175 | 177 | 352
Race/Ethnicity, Customized [Number; unit: participants]
  African | 41 | 47 | 88
  Caucasian | 161 | 164 | 325
  East Asian | 23 | 23 | 46
  Hispanic | 26 | 16 | 42
  Native American | 3 | 1 | 4
  West Asian (Indian sub-continent) | 10 | 9 | 19
  Unspecified | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Portugal | 9 | 11 | 20
  France | 13 | 14 | 27
  United States | 64 | 60 | 124
  Taiwan | 20 | 19 | 39
  Slovakia | 14 | 15 | 29
  Greece | 20 | 20 | 40
  Puerto Rico | 8 | 8 | 16
  Canada | 20 | 18 | 38
  Argentina | 32 | 30 | 62
  Brazil | 43 | 44 | 87
  Spain | 4 | 4 | 8
  Romania | 17 | 17 | 34
Brief Psychiatric Rating Scale (BPRS) Total Score [Mean (Standard Deviation); unit: Units on a scale] — BPRS is an 18-item clinician-administered scale used to assess the degree of severity of a subject's general psychopathological symptoms. Item scores range from 0 (not assessed) to 7 (extremely severe). Total Scores range from 0 to 126.
  Units on a scale | 13.61 (5.82) | 13.11 (5.29) | 13.36 (5.56)
Length of Current Schizophrenic Episode [Mean (Standard Deviation); unit: Days] — Length of episodes of clinical worsening of schizophrenia symptoms such that hospitalization or an increased level of care surrounding the episode was required. Increased level of care could include the addition of or change to any of the following from a lower level of care: day hospital program; outpatient crisis management; short-term psychiatric treatment in an emergency room; or an addition, increase, or switch of medication.
  Days | 179.16 (152.58) | 170.73 (143.34) | 174.98 (147.98)
Age of Onset of Illness [Mean (Standard Deviation); unit: Years] | 25.95 (9.21) | 26.52 (8.65) | 26.24 (8.93)
Number of Schizophrenic Episodes or Exacerbations in the Previous 24 Months [Mean (Standard Deviation); unit: Episodes] — Number of episodes of clinical worsening of schizophrenia symptoms such that hospitalization or an increased level of care surrounding the episode was required. Increased level of care could include the addition of or change to any of the following from a lower level of care: day hospital program; outpatient crisis management; short-term psychiatric treatment in an emergency room; or an addition, increase, or switch of medication.
  Episodes | 2.78 (1.81) | 2.67 (1.43) | 2.73 (1.63)
Positivie and Negative Syndrome Scale (PANSS) Scores [Mean (Standard Deviation); unit: Units on a scale] — Assesses the positive symptoms, negative symptoms, and general psychopathology specifically associated with schizophrenia. The scale consists of 30 items. Each item is rated on a scale from 1 (symptom not present) to 7 (symptoms extremely severe). Scores for PANSS positive and negative each range from 7 to 49. Scores for General Psychopathology range from 16 to 112. The sum of all 30 items is defined as the PANSS total score and ranges from 30 to 210.
  Units on a scale
    PANSS Total | 56.78 (9.76) | 56.50 (8.70) | 56.64 (9.24)
    PANSS Positive | 12.93 (3.62) | 12.40 (3.33) | 12.67 (3.49)
    PANSS Negative | 15.84 (4.23) | 16.28 (3.93) | 16.06 (4.08)
    PANSS General Pathology | 28.00 (5.45) | 27.81 (4.92) | 27.91 (5.19)
Clinical Global Impressions of Severity (CGI-S) [Mean (Standard Deviation); unit: Units on a scale] — CGI-S measures severity of illness at baseline. Scores range from 1 (normal, not at all ill) to 7 (among the most extremely ill patients).
  Units on a scale | 3.24 (0.77) | 3.26 (0.66) | 3.25 (0.72)

OUTCOME MEASURES:

1. Primary Outcome: Median Time to Discontinuation for Any Reason (Excluding Sponsor Decision)
Time Frame: Baseline up to 104 weeks
Population: All data was analyzed on an intent-to-treat (ITT) basis. An ITT analysis is an analysis of all randomized patients, with patients allocated to the treatment to which they were randomized even if a patient does not take the assigned treatment, does not receive the correct treatment, or otherwise does not follow the protocol.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Olanzapine Pamoate Depot | Oral Olanzapine
Number analyzed (Participants) | 264 | 260
Days | 644.50 [162.00 to 740.00] | 677.50 [169.50 to 740.00]
Statistical Analysis 1: Comparison: Olanzapine Pamoate Depot vs Oral Olanzapine; Test type: Superiority or Other; p = 0.612, Log Rank

2. Secondary Outcome: Change From Baseline in Heinrich-Carpenter Quality of Life in Schizophrenia Scale (QLS) Total Score at 104 Weeks
Description: Interviewer-rated scale which measures the impact of negative symptoms on occupational, social, and psychological functioning in patients with schizophrenia or schizoaffective disorder. Each of 21 items is rated on a scale from 0 (severely impaired functioning) to 6 (normal or adequate functioning). Total score range is 0-126. Least Squares Mean (LS Mean) values were adjusted for investigator and treatment at baseline, and the change values were also adjusted for baseline.
Time Frame: Baseline, 104 weeks
Population: All data were analyzed on ITT basis. ITT analysis: analysis of all randomized patients allocated to the randomized treatment even if they did not take assigned treatment, did not receive correct treatment, or otherwise did not follow the protocol. Assessment of baseline-to-endpoint change based on mixed-model repeated measures (MMRM) methodology.
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | Olanzapine Pamoate Depot | Oral Olanzapine
Number analyzed (Participants) | 130 | 135
Units on a Scale
  Baseline (n=193,193) | 60.09 (1.79) | 57.73 (1.80)
  Change from Baseline at Week 104 (n=130,135) | 8.15 (1.57) | 7.24 (1.56)
Statistical Analysis 1: Comparison: Olanzapine Pamoate Depot vs Oral Olanzapine; Test type: Superiority or Other; p = 0.649, ANCOVA — P-Value is for change from baseline at Week 104; Model: Change = Therapy, Investigator, Visit, Therapy*Visit Baseline

3. Secondary Outcome: Change From Baseline in 36-Item Short Form Health Survey (SF-36) at 104 Weeks, All Domains and Summary Scores
Description: SF-36 Health Status Survey is a generic, health-related scale assessing subjects' quality of life on 8 domains. Domains and scores: general health=5-25; physical functioning=10-30; role-physical=4-8; role-emotional=3-6; social functioning=2-10; bodily pain=2-11; vitality=4-24; mental health=5-30. There are 2 summary scores (mental component summary [MCS] and physical component summary [PCS]). MCS and PCS scores=0-100 (higher scores indicate better health status). LS Mean values were adjusted for investigator and treatment at baseline; change values were also adjusted for baseline.
Time Frame: Baseline, 104 weeks
Population: All data analyzed on ITT basis. ITT analysis: analysis of all randomized patients with patients allocated to the treatment to which they were randomized even if they did not take assigned treatment, did not receive the correct treatment, or otherwise did not follow the protocol. Assessment of baseline-to-endpoint change based on MMRM methodology.
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | Olanzapine Pamoate Depot | Oral Olanzapine
Number analyzed (Participants) | 131 | 134
Units on a Scale
  Mental Score Detail at Baseline (n=188,193) | 42.12 (1.02) | 40.56 (1.01)
  Mental Score Detail Change at Week 104 (n=124,134) | 4.87 (0.89) | 4.52 (0.87)
  Physical Score Detail at Baseline (n=188,193) | 47.80 (0.73) | 47.91 (0.72)
  Physical Score Detail Change Week 104 (n=124,134) | 0.43 (0.75) | 0.84 (0.73)
  Physical Functioning at Baseline (n=193,194) | 76.18 (2.02) | 75.63 (2.03)
  Physical Functioning Change Week 104 (n=129,134) | 1.35 (1.89) | 2.44 (1.87)
  Role-Physical at Baseline (n=192,194) | 63.60 (3.42) | 60.74 (3.43)
  Role-Physical Change at Week 104 (n=130,134) | 10.70 (3.42) | 13.76 (3.38)
  Mental Health at Baseline (n=192,194) | 61.18 (1.84) | 60.10 (1.83)
  Mental Health Change at Week 104 (n=129,134) | 5.81 (1.59) | 5.27 (1.57)
  Bodily Pain at Baseline (n=193,194) | 73.13 (2.21) | 75.61 (2.23)
  Bodily Pain Change at Week 104 (n=131,134) | 3.23 (2.12) | -0.60 (2.10)
  General Health at Baseline (n=191,194) | 60.50 (1.73) | 59.57 (1.73)
  General Health Change at Week 104 (n=128,134) | 2.69 (1.80) | 5.32 (1.77)
  Social Functioning at Baseline (n=193,194) | 64.02 (2.24) | 62.61 (2.25)
  Social Functioning Change at Week 104 (n=131,134) | 8.13 (2.18) | 5.10 (2.16)
  Vitality at Baseline (n=193,194) | 54.07 (1.81) | 49.67 (1.82)
  Vitality Change at Week 104 (n=129,134) | 7.95 (1.67) | 9.01 (1.66)
  Role-Emotional at Baseline (n=191,193) | 61.45 (3.60) | 55.34 (3.59)
  Role-Emotional Change at Week 104 (n=129,134) | 16.38 (3.54) | 17.59 (3.49)
Statistical Analysis 1: Comparison: Olanzapine Pamoate Depot vs Oral Olanzapine; Test type: Superiority or Other; p = 0.744, ANCOVA — P-value for change at Week 104 in Mental Score Detail; Change = Therapy, Investigator, Visit, Therapy*Visit, Baseline
Statistical Analysis 2: Comparison: Olanzapine Pamoate Depot vs Oral Olanzapine; Test type: Superiority or Other; p = 0.653, ANCOVA — P-value for change at Week 104 in Physical Score Detail; Change = Therapy, Investigator, Visit, Therapy*Visit, Baseline
Statistical Analysis 3: Comparison: Olanzapine Pamoate Depot vs Oral Olanzapine; Test type: Superiority or Other; p = 0.640, ANCOVA — P-value for change at Week 104 in Physical Functioning; Change = Therapy, Investigator, Visit, Therapy*Visit, Baseline
Statistical Analysis 4: Comparison: Olanzapine Pamoate Depot vs Oral Olanzapine; Test type: Superiority or Other; p = 0.454, ANCOVA — P-value for change at Week 104 in Role-Physical; Change = Therapy, Investigator, Visit, Therapy*Visit, Baseline
Statistical Analysis 5: Comparison: Olanzapine Pamoate Depot vs Oral Olanzapine; Test type: Superiority or Other; p = 0.135, ANCOVA — P-value for change at Week 104 in Bodily Pain; Change = Therapy, Investigator, Visit, Therapy*Visit, Baseline
Statistical Analysis 6: Comparison: Olanzapine Pamoate Depot vs Oral Olanzapine; Test type: Superiority or Other; p = 0.229, ANCOVA — P-value for change at Week 104 in General Health; Change = Therapy, Investigator, Visit, Therapy*Visit, Baseline
Statistical Analysis 7: Comparison: Olanzapine Pamoate Depot vs Oral Olanzapine; Test type: Superiority or Other; p = 0.594, ANCOVA — P-value for change at Week 104 in Vitality; Change = Therapy, Investigator, Visit, Therapy*Visit, Baseline
Statistical Analysis 8: Comparison: Olanzapine Pamoate Depot vs Oral Olanzapine; Test type: Superiority or Other; p = 0.256, ANCOVA — P-value for change at Week 104 in Social Functioning; Change = Therapy, Investigator, Visit, Therapy*Visit, Baseline
Statistical Analysis 9: Comparison: Olanzapine Pamoate Depot vs Oral Olanzapine; Test type: Superiority or Other; p = 0.775, ANCOVA — P-value for change at Week 104 in Role-Emotional; Change = Therapy, Investigator, Visit, Therapy*Visit, Baseline
Statistical Analysis 10: Comparison: Olanzapine Pamoate Depot vs Oral Olanzapine; Test type: Superiority or Other; p = 0.781, ANCOVA — P-value for change at Week 104 in Mental Health; Change = Therapy, Investigator, Visit, Therapy*Visit, Baseline

4. Secondary Outcome: Change From Baseline in Overall Health Status Assessment Using the EuroQol: 5 Dimensions Questionnaire (EQ-5D) at 104 Weeks
Description: Generic, multidimensional, health-related, quality-of-life instrument. Overall health status is self-reported using a visual analogue scale marked on a scale of 0 to 100 with 0 representing worst imaginable health state and 100 representing best imaginable health state. LS Mean values were adjusted for investigator and treatment at baseline; change values were also adjusted for baseline.
Time Frame: Baseline, 104 weeks
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | Olanzapine Pamoate Depot | Oral Olanzapine
Number analyzed (Participants) | 128 | 130
Units on a Scale
  Baseline (n=193,192) | 66.51 (4.58) | 72.18 (4.66)
  Change from Baseline to Week 104 (n=128,130) | 0.07 (0.02) | 0.09 (0.02)
Statistical Analysis 1: Comparison: Olanzapine Pamoate Depot vs Oral Olanzapine; Test type: Superiority or Other; p = 0.465, ANCOVA — P-value is for change from baseline to Week 104; Change = Therapy, Investigator, Visit, Therapy*Visit, Baseline

5. Secondary Outcome: Change From Baseline in Burden Assessment Scale (BAS) Total Score at 104 Weeks
Description: Self-rated scale completed by patient's caregiver which measures level of burden placed on the caregiver by caring for the patient. Each of 19 items is rated on a scale from 0 (no impact) to 3 (high negative impact). Total Score range is 0-57. If any of the 19 questions were answered "not applicable", then a Total Score of 9 was entered. LS Mean values were adjusted for investigator and treatment at baseline, and the change values were also adjusted for baseline.
Time Frame: Baseline, 104 weeks
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | Olanzapine Pamoate Depot | Oral Olanzapine
Number analyzed (Participants) | 68 | 64
Units on a Scale
  Baseline (n=104,103) | 20.06 (1.29) | 20.90 (1.24)
  Change from Baseline to Week 104 (n=68,64) | -5.02 (1.27) | -4.14 (1.29)
Statistical Analysis 1: Comparison: Olanzapine Pamoate Depot vs Oral Olanzapine; Test type: Superiority or Other; p = 0.581, ANCOVA — P-value is for change from baseline to Week 104; Change = Therapy, Investigator, Visit, Therapy*Visit, Baseline

6. Secondary Outcome: Resource Utilization: Number of Outpatient Physician Visits During the Study
Description: Number of outpatient physician visits during the study, post-baseline through 104 weeks.
Time Frame: Baseline through 104 weeks
Population: All data was analyzed on an intent-to-treat basis. An intent-to-treat analysis is an analysis of all randomized patients, with patients allocated to the treatment to which they were randomized even if a patient does not take the assigned treatment, does not receive the correct treatment, or otherwise does not follow the protocol.
Measure: Mean (Standard Deviation); unit: Outpatient physician visits
Arm/Group | Olanzapine Pamoate Depot | Oral Olanzapine
Number analyzed (Participants) | 28 | 26
Outpatient physician visits | 0.32 (1.33) | 0.65 (1.57)

7. Secondary Outcome: Resource Utilization: Days of Unpaid Care, Days of Workdays Missed, Days of Paid Care Per Week During the Study
Description: Number of days of unpaid care, number of days of workdays missed, number of days of paid care per week during the study, post-baseline through 104 weeks.
Time Frame: Baseline through 104 weeks
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Olanzapine Pamoate Depot | Oral Olanzapine
Number analyzed (Participants) | 25 | 25
Days
  Days of unpaid care per week (n=25,25) | 1.68 (3.05) | 1.40 (2.86)
  Paid workdays missed per week (n=21,23) | 0.00 (0.00) | 0.00 (0.00)
  Days of paid care per week (n=21,23) | 0.00 (0.00) | 0.00 (0.00)

8. Secondary Outcome: Number of Hospitalization Days
Description: Mean - calculated based on total number of hospitalization days per patient within reporting interval.
Time Frame: Baseline through 104 weeks
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Olanzapine Pamoate Depot | Oral Olanzapine
Number analyzed (Participants) | 264 | 260
Days | 0.43 (1.99) | 1.80 (9.30)
Statistical Analysis 1: Comparison: Olanzapine Pamoate Depot vs Oral Olanzapine; Test type: Superiority or Other; p = 0.020, ANOVA; P-value is type III p-value of ANOVA model: Total number of hospitalization days = Therapy

9. Secondary Outcome: Change From Baseline in Scale to Assess Unawareness of Mental Disorder (SUMD) Total Score at 104 Weeks
Description: Interviewer-rated scale that assesses patients' awareness of and insight into their illness. SUMD can either be based on 4 items or 5 items. Items 1 through 4 are rated from 1 (aware) to 5 (unaware); item 5 assesses correct attribution of symptoms to a mental disorder and is rated from 1 (symptoms correctly attributed) to 5 (symptoms incorrectly attributed). Total Scores for Items (1-4) range from 4 to 20 and Total Scores for Items (1-5) range from 5 to 25. LS Mean values were adjusted for investigator and treatment at baseline, and the change values were also adjusted for baseline.
Time Frame: Baseline, 104 weeks
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | Olanzapine Pamoate Depot | Oral Olanzapine
Number analyzed (Participants) | 211 | 200
Units on a Scale
  Total Score (Items 1-5) Baseline | 11.12 (0.38) | 10.73 (0.39)
  Total Score (Items 1-5) Change to Week 104 | -0.72 (0.35) | -0.50 (0.35)
  Total Score (Items 1-4) Baseline | 8.81 (0.31) | 8.52 (0.32)
  Total Score (Items 1-4) Change to Week 104 | -0.39 (0.27) | -0.29 (0.28)
Statistical Analysis 1: Comparison: Olanzapine Pamoate Depot vs Oral Olanzapine; Test type: Superiority or Other; p = 0.583, ANCOVA — P-value is for Total Score (Items 1-5) change to Week 104; Model: change = investigator, treatment, and baseline
Statistical Analysis 2: Comparison: Olanzapine Pamoate Depot vs Oral Olanzapine; Test type: Superiority or Other; p = 0.747, ANCOVA — P-value is for Total Score (Items 1-4) change to Week 104; Model: change = investigator, treatment, and baseline

10. Secondary Outcome: Change From Baseline in Working Alliance Inventory (WAI) Total Score at 104 Weeks
Description: Self-rated scale assessing patients' level of alliance with their therapist, including agreement on goals, tasks, and emotional bond. Each of 12 items is rated from 1 ('never') to 7 ('always'), with higher scores indicating greater alliance. Total Scores range from 12-84. LS Mean values were adjusted for investigator and treatment at baseline, and the change values were also adjusted for baseline.
Time Frame: Baseline, 104 weeks
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | Olanzapine Pamoate Depot | Oral Olanzapine
Number analyzed (Participants) | 195 | 184
Units on a Scale
  Baseline | 63.83 (0.96) | 63.21 (1.02)
  Change from Baseline to Week 104 | -0.92 (0.82) | -0.07 (0.88)
Statistical Analysis 1: Comparison: Olanzapine Pamoate Depot vs Oral Olanzapine; Test type: Superiority or Other; p = 0.371, ANCOVA — P-value is for change from baseline to Week 104; Model: change = investigator, treatment, and baseline

11. Secondary Outcome: Change From Baseline in Schizophrenia Objective Functioning Instrument (SOFI) Global Score at 104 Weeks
Description: Interviewer-rated 49-item scale used to assess 4 functional domains in patients with schizophrenia : 1) living situation, 2) instrumental activities of daily living, 3) productive activities and role functioning, and 4) social/recreational functioning. Possible responses and scoring vary by item and by domain, with higher scores representing better functioning. Range of possible scores is 1-100. LS Mean values were adjusted for investigator and treatment at baseline, and the change values were also adjusted for baseline.
Time Frame: Baseline, 104 weeks
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | Olanzapine Pamoate Depot | Oral Olanzapine
Number analyzed (Participants) | 120 | 124
Units on a Scale
  Baseline | 60.68 (1.39) | 60.47 (1.44)
  Change from Baseline to Week 104 | 3.92 (1.27) | 3.26 (1.29)
Statistical Analysis 1: Comparison: Olanzapine Pamoate Depot vs Oral Olanzapine; Test type: Superiority or Other; p = 0.681, ANCOVA — P-value is fro change from baseline to Week 104; Model: Change = Therapy, Investigator, Visit, Therapy*Visit, Baseline

12. Secondary Outcome: Patient Satisfaction With Medication Questionnaire-Modified (PSMQ) at 104 Weeks (All Items)
Description: Self-rated scale which measures patient's level of satisfaction with current antipsychotic medication. Consists of 3 items assessing satisfaction with current study medication (scored from 1-'very dissatisfied' to 5-'very satisfied'), preference comparing current study medication versus previous medications (scored from 1-'much prefer previous medication' to 5-'much prefer study medication'), and side effects of current study medication compared with previous medications (scored from 1-'much less side effects' to 5-'much more side effects'). Range of possible scores is 3-15.
Time Frame: 104 weeks
Population: All data analyzed on an ITT basis. ITT analysis: analysis of all randomized patients, with patients allocated to the treatment to which they were randomized even if they did not take assigned treatment, did not receive correct treatment, or otherwise did not follow the protocol. Assessment of baseline-to-endpoint change based on MMRM methodology.
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | Olanzapine Pamoate Depot | Oral Olanzapine
Number analyzed (Participants) | 139 | 146
Units on a Scale
  Overall satisfaction with current medication | 4.20 (0.11) | 3.96 (0.11)
  Preference current/previous medication (n=139,145) | 3.68 (0.10) | 3.83 (0.10)
  Side effects - current vs previous medication | 1.91 (0.10) | 1.99 (0.10)
Statistical Analysis 1: Comparison: Olanzapine Pamoate Depot vs Oral Olanzapine; Test type: Superiority or Other; p = 0.60, ANCOVA — P-value is for overall satisfaction with current medication; Model: Actual Result = Therapy, Investigator, Visit, Therapy*Visit
Statistical Analysis 2: Comparison: Olanzapine Pamoate Depot vs Oral Olanzapine; Test type: Superiority or Other; p = .258, ANCOVA — P-value is for preference current/previous medication; Model: Actual Result = Therapy, Investigator, Visit, Therapy*Visit
Statistical Analysis 3: Comparison: Olanzapine Pamoate Depot vs Oral Olanzapine; Test type: Superiority or Other; p = 0.492, ANCOVA — P-value is for side effects - current vs previous medication; Model: Actual Result = Therapy, Investigator, Visit, Therapy*Visit

13. Secondary Outcome: Patient Attitude Toward Treatment Using the Drug Attitude Inventory (DAI) Scale Total Score at 104 Weeks
Description: Self-rated scale which measures patient's subjective feelings about taking medications. Each of 10 items is rated as true or false. For items 1, 3, 4, 6, 7, 9, and 10, true is scored as 1; false is scored as 0. For items 2, 5, and 8, true is scored as 0; false is scored as 1. Possible total scores range from 0-10. A subject who answers all 10 questions false will have a score of 3; a subject who answers all 10 questions true will have a score of 7. For 7 out of 10 questions, false is represented by 0, the other 3 questions false is represented by a value=1.
Time Frame: 104 weeks
Population: as for outcome 12
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | Olanzapine Pamoate Depot | Oral Olanzapine
Number analyzed (Participants) | 137 | 143
Units on a Scale | 7.44 (0.15) | 7.47 (0.15)
Statistical Analysis 1: Comparison: Olanzapine Pamoate Depot vs Oral Olanzapine; Test type: Superiority or Other; p = 0.854, ANCOVA; Model: Actual Result = Therapy, Investigator, Visit, Therapy*Visit

14. Secondary Outcome: Number of Participants With All-Cause Discontinuations (Excluding Sponsor Decision)
Description: Number of participants who discontinued study participation for any reason (excluding sponsor decision).
Time Frame: Baseline through 104 weeks
Population: as for outcome 6
Measure: Number; unit: Participants
Arm/Group | Olanzapine Pamoate Depot | Oral Olanzapine
Number analyzed (Participants) | 264 | 260
Participants | 142 | 133
Statistical Analysis 1: Comparison: Olanzapine Pamoate Depot vs Oral Olanzapine; Test type: Superiority or Other; p = 0.600, Fisher Exact

15. Secondary Outcome: Change From Baseline in Clinical Global Impression - Severity of Illness (CGI-S) Scale Scores at 104 Weeks
Description: Measures severity of illness at the time of assessment compared with start of treatment. Scores range from 1 (normal, not at all ill) to 7 (among the most extremely ill patients).
Time Frame: Baseline, 104 weeks
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | Olanzapine Pamoate Depot | Oral Olanzapine
Number analyzed (Participants) | 121 | 128
Units on a Scale | -0.36 (0.07) | -0.27 (0.07)
Statistical Analysis 1: Comparison: Olanzapine Pamoate Depot vs Oral Olanzapine; Test type: Superiority or Other; p = 0.282, ANCOVA; Model: Change = Therapy, Investigator, Visit, Therapy*Visit Baseline

16. Secondary Outcome: Change From Baseline in Positive and Negative Syndrome Scale (PANSS) Total and Subscale Scores at 104 Weeks
Description: Assesses the positive symptoms, negative symptoms, and general psychopathology specifically associated with schizophrenia. The scale consists of 30 items. Each item is rated on a scale from 1 (symptom not present) to 7 (symptoms extremely severe). The sum of the 30 items is defined as the PANSS total score and ranges from 30 to 210.
Time Frame: Baseline, 104 weeks
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | Olanzapine Pamoate Depot | Oral Olanzapine
Number analyzed (Participants) | 121 | 128
Units on a Scale
  PANSS Total Score | -0.82 (1.15) | -1.14 (1.15)
  PANSS Positive Score | -0.48 (0.29) | -0.42 (0.29)
  PANSS Negative Score | -0.20 (0.38) | -0.41 (0.38)
  PANSS General Psychopathology Score | -0.51 (0.57) | -0.61 (0.56)
Statistical Analysis 1: Comparison: Olanzapine Pamoate Depot vs Oral Olanzapine; Test type: Superiority or Other; p = 0.834, ANCOVA — P-value is for PANSS Total Score; Model: Change = Therapy, Investigator, Visit, Therapy*Visit Baseline
Statistical Analysis 2: Comparison: Olanzapine Pamoate Depot vs Oral Olanzapine; Test type: Superiority or Other; p = 0.871, ANCOVA — P-value is for PANSS Positive Score; Model: Change = Therapy, Investigator, Visit, Therapy*Visit Baseline
Statistical Analysis 3: Comparison: Olanzapine Pamoate Depot vs Oral Olanzapine; Test type: Superiority or Other; p = 0.692, ANCOVA — P-value is for PANSS Negative Score; Model: Change = Therapy, Investigator, Visit, Therapy*Visit, Baseline
Statistical Analysis 4: Comparison: Olanzapine Pamoate Depot vs Oral Olanzapine; Test type: Superiority or Other; p = 0.893, ANCOVA — P-value is for PANSS General Psychopathology Score; Model: Change = Therapy, Investigator, Visit, Therapy*Visit, Baseline

17. Secondary Outcome: Median Time to Relapse
Description: Relapse is defined as any 1 of the following: 1) hospitalization for symptoms related to schizophrenia; 2) increase of 25% from baseline in PANSS total score (range:30-210) (if baseline score was >40) or increase of 10 points (if baseline score was ≤40), and ≥1-point increase from baseline on CGI-S score (range:1-7), provided that increase results in CGI-S ≥4; 3) deliberate self-injury or injury to others deemed clinically to be associated with worsening of psychosis; 4) discontinuation from the study because of worsening of psychosis. On PANSS and CGI-S higher scores indicate greater illness.
Time Frame: Baseline to time of relapse (up to 104 weeks)
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Olanzapine Pamoate Depot | Oral Olanzapine
Number analyzed (Participants) | 264 | 260
Days | 539.00 [105.00 to 736.00] | 623.50 [122.00 to 736.50]
Statistical Analysis 1: Comparison: Olanzapine Pamoate Depot vs Oral Olanzapine; Test type: Superiority or Other; p = 0.585, Log Rank

18. Secondary Outcome: Number of Participants Experiencing Relapse
Description: Relapse is defined as any one of the following: 1) hospitalization for symptoms related to schizophrenia; 2) an increase of 25% from baseline in the total score on the PANSS (if the baseline score was >40), or an increase of 10 points (if baseline score was <=40) and >=1-point increase from baseline score on the CGI-S score, provided that the increase results in a CGI-S score >=4; 3) deliberate self-injury or injury to others that is deemed clinically to be associated with worsening of psychosis; 4) discontinuation from the study because of worsening of psychosis.
Time Frame: Baseline through 104 weeks
Population: as for outcome 6
Measure: Number; unit: Participants
Arm/Group | Olanzapine Pamoate Depot | Oral Olanzapine
Number analyzed (Participants) | 264 | 260
Participants | 53 | 48
Statistical Analysis 1: Comparison: Olanzapine Pamoate Depot vs Oral Olanzapine; Test type: Superiority or Other; p = 0.659, Fisher Exact

19. Secondary Outcome: Change From Baseline in Brief Psychiatric Rating Scale (BPRS) Total Score at 104 Weeks
Description: BPRS is an 18-item clinician-administered scale used to assess the degree of severity of a subject's general psychopathological symptoms. For this study, the BPRS total score was derived from 18 PANSS questions. To calculate the score, the score of the 18 questions was added then 18 was subtracted from the total. As an example, if a subject had a score=1 (absent) on all 18 items, the resulting total=zero. Responses range from 0 (absent) to 6 (extremely severe); the Total Score range is 0-108.
Time Frame: Baseline, 104 weeks
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Olanzapine Pamoate Depot | Oral Olanzapine
Number analyzed (Participants) | 121 | 128
Units on a scale | -0.96 (0.60) | -0.91 (0.60)
Statistical Analysis 1: Comparison: Olanzapine Pamoate Depot vs Oral Olanzapine; Test type: Superiority or Other; p = 0.952, ANCOVA; Model: Change = Therapy, Investigator, Visit, Therapy*Visit Baseline

20. Secondary Outcome: Resource Utilization: Number of Outpatient Surgeries During the Study, 24 Months After Randomization
Description: Number of outpatient surgeries during the study, post-baseline through 104 weeks.
Time Frame: Baseline through 104 Weeks
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Surgeries
Arm/Group | Olanzapine Pamoate Depot | Oral Olanzapine
Number analyzed (Participants) | 28 | 26
Surgeries | 0.00 (0.00) | 0.04 (0.20)

21. Secondary Outcome: Change From Baseline in Weight at 104 Weeks
Time Frame: Baseline, 104 weeks
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | Olanzapine Pamoate Depot | Oral Olanzapine
Number analyzed (Participants) | 260 | 255
Kilograms
  Baseline | 81.56 (21.06) | 79.84 (19.04)
  Change from Baseline to Week 104 | 2.04 (7.19) | 2.18 (7.33)
Statistical Analysis 1: Comparison: Olanzapine Pamoate Depot vs Oral Olanzapine; Test type: Superiority or Other; p = 0.777, ANCOVA — P-value is for change from baseline to Week 104; Model: change = baseline, treatment, and investigator

22. Secondary Outcome: Participants With Potentially Clinically Significant (PCS) Weight Gain at 104 Weeks
Description: PCS weight gain is defined as a >=7% increase in weight from baseline at 104 weeks.
Time Frame: Baseline, 104 weeks
Population: as for outcome 6
Measure: Number; unit: Participants
Arm/Group | Olanzapine Pamoate Depot | Oral Olanzapine
Number analyzed (Participants) | 260 | 255
Participants | 106 | 97
Statistical Analysis 1: Comparison: Olanzapine Pamoate Depot vs Oral Olanzapine; Test type: Superiority or Other; p = 0.530, Fisher Exact

23. Secondary Outcome: Participants With Normal to High Fasting Glucose, Fasting Total Cholesterol, and Fasting Triglycerides
Description: Normal to high fasting glucose = <100 milligrams per deciliter (mg/dL) baseline; >=126 mg/dL any time post baseline (or endpoint). Normal to high fasting total cholesterol =<200 mg/dL baseline; >=240 mg/dL any time post baseline or endpoint. Fasting triglycerides <150 mg/dL baseline; >=200 mg/dL and <500 mg/dL any time post baseline or endpoint.
Time Frame: Baseline through 104 weeks
Population: as for outcome 6
Measure: Number; unit: Participants
Arm/Group | Olanzapine Pamoate Depot | Oral Olanzapine
Number analyzed (Participants) | 243 | 241
Participants
  Fasting Glucose (n=243,241) | 25 | 17
  Fasting Total Cholesterol (n=242,231) | 12 | 14
  Fasting Triglycerides (n=242,231) | 48 | 44
Statistical Analysis 1: Comparison: Olanzapine Pamoate Depot vs Oral Olanzapine; Test type: Superiority or Other; p = 0.258, Fisher Exact — P-value for fasting glucose
Statistical Analysis 2: Comparison: Olanzapine Pamoate Depot vs Oral Olanzapine; Test type: Superiority or Other; p = 0.688, Fisher Exact — P-value is for fasting total cholesterol
Statistical Analysis 3: Comparison: Olanzapine Pamoate Depot vs Oral Olanzapine; Test type: Superiority or Other; p = 0.908, Fisher Exact — P-value is for fasting triglycerides

24. Secondary Outcome: Participants With Treatment-Emergent Abnormal High Prolactin at 104 Weeks
Description: The prolactin reference Range is: Female: 2.0 - 29.0 nanograms per milliliter (ng/mL); Male: 2.0 - 20.0 ng/mL. A treatment-emergent abnormally high value is defined as a change from a value less than or equal to the high limit at all baseline visits to a value greater than the high limit at any time after baseline.
Time Frame: Baseline, 104 weeks
Population: as for outcome 6
Measure: Number; unit: Participants
Arm/Group | Olanzapine Pamoate Depot | Oral Olanzapine
Number analyzed (Participants) | 226 | 217
Participants | 12 | 12
Statistical Analysis 1: Comparison: Olanzapine Pamoate Depot vs Oral Olanzapine; Test type: Superiority or Other; p = 0.835, Fisher Exact

25. Secondary Outcome: Participants With Treatment-Emergent High Alanine Transaminase (ALT), Aspartate Transaminase (AST), and Total Bilirubin
Description: Treatment-emergent (TE) high ALT is defined as a baseline value of <3 times the upper limit of normal (ULN) to >=3 times the ULN at endpoint. TE high AST is defined as a baseline value of <5 times the ULN to >=5 times the ULN at endpoint. TE high total bilirubin is defined as a baseline value of <2 times the ULN to >=2 times the ULN at endpoint. Hy's Rule is defined as ALT >=3 times the ULN and total bilirubin >=2 times the ULN.
Time Frame: Baseline through 104 Weeks
Population: as for outcome 6
Measure: Number; unit: Participants
Arm/Group | Olanzapine Pamoate Depot | Oral Olanzapine
Number analyzed (Participants) | 256 | 253
Participants
  ALT (n=255,251) | 11 | 12
  AST (n=256,252) | 3 | 4
  Total bilirubin (n=256,253) | 0 | 2
  Hy's Rule (n=255,251) | 0 | 0
Statistical Analysis 1: Comparison: Olanzapine Pamoate Depot vs Oral Olanzapine; Test type: Superiority or Other; p = 0.834, Fisher Exact — P-value is for ALT
Statistical Analysis 2: Comparison: Olanzapine Pamoate Depot vs Oral Olanzapine; Test type: Superiority or Other; p = 0.723, Fisher Exact — P-value is for AST
Statistical Analysis 3: Comparison: Olanzapine Pamoate Depot vs Oral Olanzapine; Test type: Superiority or Other; p = 0.247, Fisher Exact — P-value is for total bilirubin

26. Secondary Outcome: Participants Discontinuing Because of an Adverse Event (AE) or Death
Time Frame: Baseline through 104 weeks
Population: as for outcome 6
Measure: Number; unit: Participants
Arm/Group | Olanzapine Pamoate Depot | Oral Olanzapine
Number analyzed (Participants) | 264 | 260
Participants | 26 | 27
Statistical Analysis 1: Comparison: Olanzapine Pamoate Depot vs Oral Olanzapine; Test type: Superiority or Other; p = 0.885, Fisher Exact

ADVERSE EVENTS:
Arm/Group | Olanzapine Pamoate Depot | Oral Olanzapine
Serious Adverse Events (participants affected / at risk) | 25/264 | 34/260
Other Adverse Events (participants affected / at risk) | 177/264 | 165/260
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Olanzapine Pamoate Depot (N=264) | Oral Olanzapine (N=260)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1) — This event resulted in death.
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 2 (2)
Pneumonia (Infections and infestations) | 1 (1) | 3 (3)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) — This event resulted in death.
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Intentional overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Ependymoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Acute psychosis (Psychiatric disorders) | 0 (0) | 1 (1)
Aggression (Psychiatric disorders) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1)
Alcohol abuse (Psychiatric disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (2) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1)
Depressive symptom (Psychiatric disorders) | 1 (1) | 0 (0)
Hallucination, auditory (Psychiatric disorders) | 0 (0) | 1 (1)
Homicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1)
Impulsive behaviour (Psychiatric disorders) | 0 (0) | 1 (1)
Paranoia (Psychiatric disorders) | 0 (0) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 4 (4) | 3 (3)
Schizophrenia (Psychiatric disorders) | 10 (10) | 9 (9)
Suicidal ideation (Psychiatric disorders) | 2 (2) | 1 (1)
Suicide attempt (Psychiatric disorders) | 1 (1) | 3 (3)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoaesthesia facial (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Arterial thrombosis limb (Vascular disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Hypovolaemic shock (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Olanzapine Pamoate Depot (N=264) | Oral Olanzapine (N=260)
Nasopharyngitis (Infections and infestations) | 18 (23) | 14 (24)
Weight decreased (Investigations) | 15 (18) | 14 (15)
Weight increased (Investigations) | 44 (51) | 43 (47)
Increased appetite (Metabolism and nutrition disorders) | 17 (17) | 16 (16)
Headache (Nervous system disorders) | 12 (25) | 22 (36)
Somnolence (Nervous system disorders) | 23 (24) | 25 (28)
Anxiety (Psychiatric disorders) | 26 (37) | 18 (21)
Insomnia (Psychiatric disorders) | 29 (37) | 26 (33)
Hypertension (Vascular disorders) | 9 (11) | 13 (13)

LIMITATIONS AND CAVEATS:
Results for Outcome Measures 17 and 18 were corrected as a result of an identified programming error.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days